CLINICAL TRIAL: NCT00756470
Title: A Phase II Study of Neoadjuvant Lapatinib Plus Chemotherapy (Sequential FEC75 and Paclitaxel) in Women With Inflammatory Breast Cancer Whose Tumors Overexpress ErbB2 (Her2/Neu)
Brief Title: Phase II Neoadjuvant in Inflammatory Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0818
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Inflammatory Breast Cancer; IBC; ErbB2 overexpression; Lapatinib; Paclitaxel; 5-Fluorouracil; Epirubicin; Cyclophosphamide; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Lapatinib; Paclitaxel; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Lapatinib plus Chemotherapy (Experimental): Four cycles of Lapatinib and Paclitaxel followed by 4 cycles of Lapatinib plus 5-Fluorouracil, Cyclophosphamide, Epirubicin (FEC75). Cycle is 21 days.
  Lapatinib alone at 1,000 mg orally once daily for a 2-week run-in period, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each.
  1. Week 3 Paclitaxel 80 mg/m^2 weekly for 4 cycles (12 weeks) administered on Day 1, Day 8, and Day 15) of each cycle combined with Lapatinib 750 mg orally once daily.
  2. Week 15, second combination treatment consisting of Lapatinib (1,000 mg orally once daily) combined with FEC75 (5-FU 500 mg/m^2, Epirubicin 75 mg/m^2, and Cyclophosphamide 500 mg/m^2 every 3 weeks for 4 cycles).
  Interventions: Drug: Lapatinib; Drug: Paclitaxel; Drug: 5-Fluorouracil (5-FU); Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Lapatinib — 1000 mg taken by every day by mouth (PO) weeks 1 and 2; then starting day 15 for 12 weeks (weeks 3 to 14) daily 750 mg PO. Week 15, second combination treatment consisting of lapatinib (1,000 mg orally once daily) combined with FEC7.
  Other Names: Tykerb; GW572016
Drug: Paclitaxel — 80 mg/m^2 intravenously over 1 hour weekly for 4 cycles administered on Day 1, Day 8, and Day 15 of each cycle then weekly starting day 15 for 12 weeks.
  Other Names: Taxol
Drug: 5-Fluorouracil (5-FU) — 500 mg/m^2 intravenously over 3-5 minutes every three weeks of Weeks 13-24.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Epirubicin — 75 mg/m^2 intravenously over 5-10 minutes every three weeks of Weeks 13-24.
Drug: Cyclophosphamide — 500 mg/m^2 intravenously over 45-60 minutes every three weeks of Weeks 13-24.
  Other Names: Cytoxan; Neosar

SUMMARY:
The goal of this clinical research study is to learn how well lapatinib taken alone, followed by taking lapatinib with paclitaxel, and then taking lapatinib with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC75) works to help to control Inflammatory Breast Cancer (IBC). The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Lapatinib is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the Her2/neu receptor and the epidermal growth factor (EGFR).

Cyclophosphamide, paclitaxel, and 5-fluorouracil are designed to block cancer cells from dividing, which may slow or stop their growth and their ability to spread throughout the body. This may cause the cancer cells to die.

Epirubicin is designed to attach to DNA (the genetic material of cells) which may slow or stop their growth and cause them to die.

Study Drug Administration:

On Weeks 1-24 you will take lapatinib every day by mouth with water (about 8 ounces). It should be taken at least 1 hour before or at least 2 hours after eating. It is important that you take the study drug at about the same time every day. You should not eat pamelo fruit, grapefruit, star fruit, pawpaw, and/or drink their juices while on study.

If you forget to take a dose of the study drug, you should take the missed dose as soon as you remember, unless it has been more than 12 hours. If it has been more than 12 hours, do not take the missed dose. Instead, take the next dose as scheduled the next day. If you vomit after taking the study drug, wait until the next day to take your next dose.

The study drug should be stored at room temperature and out of direct sunlight. The study drug should be kept away from children. About every 3 weeks, you will need to bring back your empty or partially used bottle of study drug as instructed by your doctor.

On Weeks 3-12, you will receive paclitaxel through a needle in your vein 1 time a week. The infusion will take about 1 hour. You will continue to take lapatinib every day.

On Weeks 13-24, you will receive 5-fluorouracil, epirubicin, and cyclophosphamide 1 time every 21 day study cycle. You will receive 4 cycles. Each 5-fluorouracil infusion will take about 3-5 minutes, each epirubicin infusion will take about 5-10 minutes, and the cyclophosphamide infusion will take about 45-60 minutes. You will continue to take lapatinib every day during Weeks 13-24.

If you experience intolerable side effects, the study doctor may give you drugs to help with this side effect or change your dose of study drug.

Study Visits:

On Day 1 of Week 1, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any drugs that you may be taking.
* You will have a performance status evaluation.

Every 3 weeks while taking combination chemotherapy and study drug, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any changes in your health and any drugs that you may be taking.
* You will have a performance status evaluation.
* Your medical history will be recorded.
* Blood (about 3 tablespoons) will be drawn for routine tests.

At Week 6, you will have a CT scan, MRI, and/or a bone scan to check the status of the disease.

At the end of the chemotherapy treatment, the disease will be measured by physical exam, chest CT scan and sonogram to check the status of the disease. If the disease has gotten worse, you will be taken off study. If the disease has gotten worse, you will be taken off study. Your doctor will discuss your next step of treatment options.

Surgery:

At the end of the chemotherapy period, if the disease has responded well to the drugs, you will have surgery to remove the breast tumor. You will sign a separate consent form for the surgery. Either at the end-of-treatment visit at week 24 after you are done with chemotherapy, or before the surgery, the following tests will be performed:

* You will have a complete physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* You will be asked about any drugs you may be taking.
* Blood (about 3 tablespoons) will be drawn for routine tests
* You will have an ECG.
* You will have a multiple gated acquisition scan (MUGA) or echocardiogram to check your hearts health.
* You will have a CT scan, MRI, and/or a bone scan to check the status of the disease.
* You will have a tissue biopsy to check the status of the disease.

Length of Study:

You may continue to receive the study drugs for up to 24 weeks. You will be taken off study early if the disease gets worse or intolerable side effects occur.

Long-Term Follow-Up:

Once you are off study, you will have follow-up visits at 3 and 6 months after surgery. At these visits, you will have a MUGA or ECHO performed.

You will have additional visits every 4 months for Years 2 and 3, and then every 6 months for Years 4 and 5. At these visits, blood (about 3 tablespoons) will be drawn for routine tests.

This is an investigational study. Lapatinib is FDA approved and commercially available when taken in combination with capecitabine for another type of breast cancer. Using Lapatinib in inflammatory breast cancer is investigational.

5-fluorouracil, epirubicin, cyclophosphamide, and paclitaxel are all FDA approved and commercially available for treating breast cancer. The combination of these drugs is not currently FDA approved for the treatment of IBC. At this time, this drug combination is only being used in research.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed informed consent form (ICF) and a Patient Authorization Form (HIPAA).
2. Histological confirmation of breast carcinoma with a clinical diagnosis of IBC based on the presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass, involving the majority of the skin of the breast. Pathologic evidence of dermal lymphatic invasion should be noted but is not required for diagnosis.
3. Tumors that overexpress ErbB2, defined as one of the following definitions: 3+ staining by immunohistochemistry and/or a FISH ratio of more than 2.2
4. Have either measurable or clinically evaluable skin disease. Patients with metastasis but are candidates for mastectomy are eligible.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 - 1.
6. Have left ventricular ejection fraction (LVEF) within the institutional range of normal as measured by either echocardiogram (ECHO) or MUGA scans. The same modality must be used consistently throughout the study.
7. Willing to under go 1 mandatory core biopsy (up to 4 passes) and 1 mandatory skin biopsy to confirm IBC diagnosis and for biologic expression profiling.Subjects with clinically palpable residual disease may undergo an optional 2nd and 3rd core needle biopsy (1 after initial 2-week Lapatinib therapy and 1 after 6 months of completing all chemotherapy, before surgery) to allow identification of presumed pathways of therapy resistance. Information may give subject options for other targeted therapies (e.g. trastuzumab) if definitive surgery confirms residual disease.
8. Are able to swallow and retain oral medication (intact pill).
9. Are able to complete all screening assessments as outlined in the protocol.
10. Have adequate organ function.
11. Are subjects aged >/= 18 years with any menopausal status: Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal) Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhea (severe), women who are perimenopausal, and young women who have begun to menstruate. Criterion continued in #13
12. These subjects must have a negative serum pregnancy test at screening and agree to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or Consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; Criterion continued in # 13
13. Any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progestogen only) where not contraindicated for this subject population or per local practice.; or barrier methods, including diaphragm or condom with a spermicide. Please note that breast cancer subjects on this trial cannot receive injectable levonorgestrel or injectable progestogen due to the potential for an adverse effect of anti-hormonal therapies on chemotherapy administered for breast cancer.

Exclusion Criteria:

1. Have received any prior to chemotherapy.
2. Had prior therapy with an ErbB1 and/or ErbB2 inhibitor.
3. Are receiving concurrent anti-cancer therapy (chemotherapy, immunotherapy, and biologic therapy) while taking study medication.
4. Have Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Women with ulcerative colitis are also excluded.
5. Have a concurrent disease or condition that would make the woman inappropriate for study participation, or any serious medical disorder that would interfere with the woman's safety.
6. Have an active or uncontrolled infection.
7. Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
8. Have active cardiac disease, defined as one or more of the following: history of uncontrolled of symptomatic angina, history of arrhythmias requiring medications, or clinically significant; myocardial infarction < 6 months from study entry; uncontrolled or symptomatic congestive heart failure; ejection fraction below the institutional normal limit; any other cardiac condition, which is in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
9. Are pregnant or breastfeeding.
10. Have received concurrent treatment with an investigational agent clinical trial.
11. Use of any prohibited medications concurrently with lapatinib therapy.
12. Have used investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.
13. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the agents used in this study or their excipients.
14. Are receiving therapeutic anti-coagulation therapy (i.e. warfarin, heparin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alvarez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 9, 2008 to December 30, 2011. All recruitment done at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow enrollment and review of futility.
Groups:
- Neoadjuvant Lapatinib Plus Chemotherapy: Four cycles of Lapatinib and Paclitaxel followed by 4 cycles of Lapatinib plus 5-Fluorouracil (5FU), Cyclophosphamide, Epirubicin (FEC75). Cycle is 21 days.
  Lapatinib alone at 1,000 mg orally once daily for a 2-week run-in period, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each.
  1. Week 3 Paclitaxel 80 mg/m^2 weekly for 4 cycles (12 weeks) administered on Day 1, Day 8, and Day 15) of each cycle combined with Lapatinib 750 mg orally once daily.
  2. Week 15, second combination treatment consisting of Lapatinib (1,000 mg orally once daily) combined with FEC75 (5-FU 500 mg/m2, epirubicin 75 mg/m^2, and Cyclophosphamide 500 mg/m^2 every 3 weeks for 4 cycles).
Period: Overall Study
Arm/Group | Neoadjuvant Lapatinib Plus Chemotherapy
Started | 15
Completed | 10
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- Neoadjuvant Lapatinib Plus Chemotherapy: Four cycles of Lapatinib and Paclitaxel followed by 4 cycles of Lapatinib plus 5-Fluorouracil, Cyclophosphamide, Epirubicin (FEC75). Cycle is 21 days.
  Lapatinib alone at 1,000 mg orally once daily for a 2-week run-in period, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each.
  1. Week 3 Paclitaxel 80 mg/m^2 weekly for 4 cycles (12 weeks) administered on Day 1, Day 8, and Day 15) of each cycle combined with Lapatinib 750 mg orally once daily.
  2. Week 15, second combination treatment consisting of Lapatinib (1,000 mg orally once daily) combined with FEC75 (5-FU 500 mg/m2, epirubicin 75 mg/m^2, and Cyclophosphamide 500 mg/m^2 every 3 weeks for 4 cycles).
Arm/Group | Neoadjuvant Lapatinib Plus Chemotherapy
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 53.8 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
ECOG (Performance Status) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status (PS) performed at baseline. PS described as 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; etc.
  participants
    PS 0 | 13
    PS 1 | 2
Clinical Stage: American Joint Committee on Cancer (AJCC) 2009 [Number; unit: participants] — AJCC Breast cancer staging: Anatomic stage 0, IA or B, IIA or B, IIIA to C or IV. AJCC staging system provides strategy for grouping participants by prognosis, based on the extent of the tumor (T), the extent of spread to the lymph nodes (N), and the presence of metastasis (M). Once the T, N, and M are determined, they are combined , and an overall stage of 0, I, II, III, IV is assigned from least advanced to more advanced. Sometimes these stages are subdivided as well, using letters such as IIIA and IIIB.
  participants
    III B | 3
    III C | 8
    IV | 4

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With pCR After Completion of All Protocol Specified Therapy & Surgery (Surgical Population)
Description: Pathologic complete response [pCR or RCB Class 0] defined as no residual invasive disease (malignant cells) in the breast or axillary lymph nodes as assessed at the time of surgery following completion of all protocol specified neoadjuvant chemotherapy, which is approximately 26 weeks following the start of neoadjuvant chemotherapy and surgery. the residual cancer burden (RCB) was estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes. The calculated RCB index value is categorized as one of four RCB classes, RCB-0 to RCB-III where RCB-0 is best prognosis (no residual disease) to RCB-III a worst prognosis. The RCB score for participants was assessed following completion of all protocol specified therapy, 4 cycles of lapatinib and paclitaxel followed by 4 cycles of lapatinib plus FEC75 and surgery.
Time Frame: Following definitive surgery at completion of neoadjuvant chemotherapy (following approximately 26 treatment weeks)
Population: While analyses was based on intent-to-treat (ITT) the surgical population includes only subjects who underwent definitive surgery (10 participants had a modified radical mastectomy) thus 5 were not evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Lapatinib Plus Chemotherapy
Number analyzed (Participants) | 10
participants
  RCB Class 0 (pCR) | 1
  RCB Class I | 0
  RCB Class II | 9
  RCB Class III | 0

2. Primary Outcome: Rate of Pathologic Complete Response (pCR) Following Neoadjuvant Chemotherapy
Description: Pathologic complete response (pCR) rate defined as number of participants out of total that had no residual invasive disease (malignant cells) in the breast or axillary lymph nodes as assessed at the time of surgery following completion of all protocol specified neoadjuvant chemotherapy, which is approximately 26 weeks following the start of neoadjuvant chemotherapy.
Time Frame: Assessed at time of surgery following completion neoadjuvant chemotherapy (approximately 26 weeks)
Population: With an intent-to-treat population analysis, all participants who received any treatment were included in the analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Neoadjuvant Lapatinib Plus Chemotherapy
Number analyzed (Participants) | 15
Percentage of Participants | 6.6

ADVERSE EVENTS:
Time Frame: Adverse event collection approximately 26 weeks following the start of neoadjuvant chemotherapy. Overall study period: October 2008 to September 2013.
Arm/Group | Neoadjuvant Lapatinib Plus Chemotherapy
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Lapatinib Plus Chemotherapy (N=15)
Diarrhea (Gastrointestinal disorders) | 7 — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 3 — Grade 3
Neutropenic Fever (Blood and lymphatic system disorders) | 1 — Grade 3
Skin Rash (Skin and subcutaneous tissue disorders) | 3 — Grade 3
Fatigue (General disorders) | 3 — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Lapatinib Plus Chemotherapy (N=15)
Anemia (Blood and lymphatic system disorders) | 2 — Grade 2
Neutropenia (Blood and lymphatic system disorders) | 2 — Grade 2
Skin Rash (Skin and subcutaneous tissue disorders) | 5 — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 — Grade 2
Liver dysfunction (Hepatobiliary disorders) | 3 — Grade 2
Decreased Ejection Fraction (Cardiac disorders) | 1 — Grade 2
Fatigue (General disorders) | 7 — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes